CLINICAL TRIAL: NCT01057914
Title: Effects of Six Months Treatment With Nutritional Supplements or Dietary Advice, Alone or in Combination on Mortality, Health-related Quality of Life and Health-care Consumption for Elderly Patients at Risk of Malnutrition.
Brief Title: Effects of Nutritional Supplementation and Dietary Advice in Elderly Patients After Hospital Discharge.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Västmanland County Council, Sweden (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: LTV-69151
Record Dates: First submitted 2010-01-27; First posted 2010-01-28 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Malnutrition
Keywords: Randomized controlled trial; Malnutrition; Aged; Aged 80 and over; Nutrition therapy
MeSH Terms: conditions — Malnutrition | interventions — Dietary Supplements; Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Supplemention (Experimental)
  Interventions: Dietary Supplement: Nutritional supplementation with a liquid formula
- Dietary advice (Experimental)
  Interventions: Other: Dietary advice
- Combination treatment (Experimental)
  Interventions: Other: Combination of supplement and dietary advice
- Usual care (No Intervention)

INTERVENTIONS:
Dietary Supplement: Nutritional supplementation with a liquid formula — The patient consumes 400 kcal from a liquid supplementation formula
  Arms: Supplemention
Other: Dietary advice — The patient receives dietary advice for one hour during the hospital stay.
  Arms: Dietary advice
Other: Combination of supplement and dietary advice — The patient receives dietary advice for one hour during the hospital stay and consumes 400 kcal from liquid supplementation formula for six month after discharge.
  Arms: Combination treatment

SUMMARY:
The purpose of this study is to evaluate the effects of nutritional therapy in elderly malnourished patients. The hypothesises are that nutritional supplementation and dietary advice alone or in combination affects mortality, quality of life and health-care consumption after six month of treatment.

ELIGIBILITY:
Inclusion Criteria:

* ≥65 years old
* Admitted to one of the participating wards during the recruitment period

Exclusion Criteria:

* Well-nourished
* No consent to participate
* Not able to communicate
* Not able to understand swedish
* Presumed life-expectancy <1 year
* Already receiving nutritional therapy including dietary advice, supplements, tube-feeding or parenteral nutrition
* Dietary restrictions due to illness or disease inconsistent with the intervention
* Impaired cognitive function or dementia
* Body mass index ≥35
* Living in old peoples homes, sheltered housing, institution, service flats or nursing homes
* Participant in a study evaluating differences in 3-year mortality between well-nourished patients, patients at risk of malnutrition and malnourished patients

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 671 (Actual)
Dates: Start 2010-02; Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
All cause mortality | Six months, one year, three years

SECONDARY OUTCOMES:
Health-related quality of life | Six months, one year, three years
Health-care consumption | Six months, one year, three years
Function in activities in daily life | Six months, one year, three years

CONTACTS AND LOCATIONS:
Overall Officials: Leif Bergkvist, Principal Investigator — Centre for clinical research, Landstinget Västmanland/Uppsala University
Locations (5):
- Sweden (5):
  - Falu lasarett, Falun, Dalarna County
  - Mälarsjukhuset in Eskilstuna, Eskilstuna, Sörmland
  - Nyköpings lasarett, Nyköping, Sörmland
  - Akademiska sjukhuset, Uppsala, Uppland
  - Västmanlands sjukhus Västerås, Västerås, Västmanland County

REFERENCES:
- [Derived] Soderstrom L, Rosenblad A, Bergkvist L, Frid H, Thors Adolfsson E. Dietary advice and oral nutritional supplements do not increase survival in older malnourished adults: a multicentre randomised controlled trial. Ups J Med Sci. 2020 Aug;125(3):240-249. doi: 10.1080/03009734.2020.1751752. Epub 2020 May 2. PMID 32362168